CLINICAL TRIAL: NCT00402961
Title: A Phase II Randomized Controlled Trial of Acupuncture for Reduction of Post-Colectomy Ileus
Brief Title: Trial of Acupuncture for Reduction of Post-Colectomy Ileus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-145; NCT00425412 (obsolete NCT alias)
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Ileus; Colon Cancer; Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: Acupuncture; Post-Colectomy Ileus; Abdominal Surgery; Colon Surgery
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Acupuncture Therapy

ARMS (2):
- 1 (Active Comparator): Acupuncture is the insertion of needles at certain body points.
  Interventions: Other: Acupuncture
- 2 (Sham Comparator): sham acupuncture
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture will be given twice daily for a total of three days (Day 1 to 3). The two acupuncture sessions will be separated by at least 4 hours, preferably given in the morning and late afternoon. Each session will last approximately 30 minutes, starting from the moment the first needle is inserted and ending the moment the first needle is removed. The last treatment will be given at the end of Day 3 or day of discharge.
  Arms: 1
Other: Sham Acupuncture — Sham Acupuncture involves the acupuncturist tapping a plastic guiding tube on the surface of the true points to produce some discernible sensation and then immediately tapping a real needle sideways parallel to the skin surface without needle insertion. It will be given twice daily for a total of three days (Day 1 to 3). The two acupuncture sessions will be separated by at least 4 hours, preferably given in the morning and late afternoon. Each session will last approximately 30 minutes, starting from the moment the first needle is inserted and ending the moment the first needle is removed. The last treatment will be given at the end of Day 3 or day of discharge,
  Arms: 2

SUMMARY:
The purpose of this study is to see whether acupuncture may help patients recover from colon cancer surgery.

DETAILED DESCRIPTION:
* To determine whether a Phase III trial of acupuncture for postoperative recovery after colorectal surgery is warranted as defined by evidence of reduction of postoperative ileus when compared to sham acupuncture.
* To explore whether acupuncture reduces the length of hospital stay more than sham acupuncture
* To explore whether acupuncture improves patient satisfaction with the hospital experience by ameliorating other postoperative symptoms such as pain and nausea and vomiting.
* To determine the feasibility of a Phase III trial in terms of sample size, accrual rate, attrition rate and data completion.

Postoperative ileus contributes to prolonged hospital stay, readmission and postoperative morbidities in patients undergoing major abdominal surgery. Reduction of postoperative ileus is important in postoperative recovery. Postoperative pain may require opioids, which further reduce gastrointestinal (GI) motility. Postoperative nausea and vomiting hamper the resumption of oral intake. Together, these three common postoperative problems contribute to patient discomfort, delayed discharge and increased overall hospitalization costs, despite current multi-modal management options. Any safe and effective therapy in addition to current standard of care would be welcomed by patients, surgeons and hospitals.

Acupuncture is a complementary medicine modality shown to reduce postoperative pain, suppress nausea and vomiting, and promote GI motility. It is associated with few adverse events. Here we propose a randomized, sham controlled phase II study to evaluate acupuncture, in addition to conventional therapy, for its safety and effectiveness in improving postoperative recovery of colorectal cancer patients undergoing segmental or subtotal colectomy. The overall objective of this developmental project is to determine whether a more extended research project is warranted.

The specific aims are:

* To determine whether a Phase III trial of acupuncture for postoperative recovery after colorectal surgery is warranted as defined by evidence for a reduction of postoperative ileus when compared to sham acupuncture. Hypothesis: acupuncture promotes upper and lower GI motility in patients experiencing postoperative ileus after colectomy more than sham acupuncture.
* To explore whether acupuncture improves patient satisfaction with the hospital experience by ameliorating other postoperative symptoms such as pain and nausea and vomiting. Hypothesis 2a: acupuncture reduces postoperative pain more than placebo in colectomy patients; 2b: acupuncture reduces postoperative nausea and vomiting more than placebo in colectomy patients.
* To determine the feasibility of a phase III trial in terms of sample size, accrual rate, attrition rate and data completion. Hypothesis 3: a phase III study of acupuncture in the treatment of post-colectomy ileus in cancer patients is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of any ethnicity
* Age over 18 years (children are not included because colorectal cancer is rare in children).
* Scheduled to undergo elective resection of biopsy proven colorectal cancer or suspected colorectal cancer

Exclusion Criteria:

Pre-operative factors:

* History of major abdominal or pelvic surgery that have caused significant alteration in anatomy and function of the GI tract which may affect the endpoints of this study.
* Laparoscopic procedures. They tend to result in less postoperative ileus.
* Administration of epidural anesthetics or epidural opioids: these have previously been shown to affect postoperative GI motility. They made up only 5% of colectomy patients in the investigators' institution.
* Acupuncture within the last 4 weeks (to exclude any possible residual effect from acupuncture)
* Contraindications to use of electrical stimulation, including cardiac pacemaker and implantable cardioverter defibrillator (ICD)
* Prior serious adverse event with acupuncture
* Intra-operative events (these events alter the postoperative recovery course significantly):

  * Resection incorporating the upper GI tract. Such surgeries are usually more complex, involving more organs and are associated with a more diverse postoperative course, making the study population more heterogeneous.
  * Gross fecal spillage (high complication rate in this setting)
  * Need to leave nasogastric tube in (contaminating the primary endpoint)
  * Decision to give epidural anesthetics or epidural opioids postoperatively (shown previously to change the major endpoints)
  * Complications during surgery requiring a patient to be transferred to the Intensive Care Unit (ICU) directly from the Operating Room or Post Anesthesia Care Unit (PACU) as this also alters the postoperative course significantly. Patients transferred to the floor first will not be excluded. They will be fully registered and randomized. If they deteriorate later during the hospital stay, requiring a transfer to the ICU, they will still be followed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine whether a Phase III trial of acupuncture for postoperative recovery after colorectal surgery is warranted as defined by evidence of reduction of postoperative ileus when compared to sham acupuncture | end of study

SECONDARY OUTCOMES:
To explore whether acupuncture improves patient satisfaction with the hospital experience by ameliorating other postoperative symptoms such as pain and nausea and vomiting | daily pain score, opioids consumption (total dose of morphine equivalent during hospitalization and average dose per day) severity of nausea as defined by number of request for PRNantiemetics, and number of emetic episodes during hospital stay.
To determine the feasibility of a Phase III trial in terms of sample size, accrual rate, attrition rate and data completion | end of study
GI-2, (also representing time to recovery of gastrointestinal [GI] function) | patient first tolerated solid food,and time patient first passed a bowel movement
GI contractions measured with a multifunctional stethoscope | duration of two minute before and immediately after each true or sham acupuncture treatment.
Daily pain score | daily during hospitalization
Opioid consumption (total dose of morphine equivalent during hospitalization and average dose per day) | daily pain score, opioids consumption (total dose of morphine equivalent during hospitalization and average dose per day) severity of nausea as defined by number of request for PRNantiemetics, and number of emetic episodes during hospital stay.
Number of emetic episodes during hospital stay | assement daily

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org